CLINICAL TRIAL: NCT04793178
Title: The Effectivity of End-tidal CO2 and Oxygen Reserve Index (ORI) Monitoring to Detect Respiratory Events and Hypoxemia Before Pulse Oxymetry in Sedation
Brief Title: The Effectivity of End-tidal CO2 and Oxygen Reserve Index (ORI) Monitoring in Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas Hospital (Other)
Responsible Party: Principal Investigator, Seyhan Yagar, Associated Professor, Yuksek Ihtisas Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: YuksekIhtisasH
Record Dates: First submitted 2017-01-23; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Hypoxemia; Procedural Sedation; Hypercapnia; Apnea
Keywords: sedation, end-tidal carbon dioxide, oxygen reserve index
MeSH Terms: conditions — Hypoxia; Hypercapnia; Apnea

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and assessor are blinded to study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen Reserve Index Blinded Group (Active Comparator): Aneshesist will be blinded for oxygen reserve index monitoring (ORI, Masimo Corporation), but he will be allowed to use pulse oxymetry and end-tidal carbon dioxide monitoring to manage the respiratory conditions and depth of sedation.
  Interventions: Device: Oxygen Reserve Index, Masimo Corporation, USA.
- Oxygen Reserve Index Group (Experimental): Aneshesist will be allowed to use pulse oxymetry, end-tidal carbon dioxide and oxygen reserve index (ORI) monitoring. He will manage the depth of sedation, respiaratory conditions.
  Interventions: Device: Oxygen Reserve Index, Masimo Corporation, USA.

INTERVENTIONS:
Device: Oxygen Reserve Index, Masimo Corporation, USA. — The oxygen reserve index (ORI) is a new feature of multiple wavelength pulse oximetry that provides real-time visibility to oxygenation status in the moderate hyperoxic range (PaO2 of approximately 100-200 mm Hg).

SUMMARY:
Endoscopic procedures are commonly performed using sedation. As drug-induced respiratory depression is a major cause of sedation-related morbidity, pulse oximetry has been established as standart practice . However SpO2 does not completely reflect ventilation. Capnography is an additional monitoring parameter which demonstrates respiration activity breath by breath. Unfortunately, in the state of moderate or deep sedation during diagnostic or therapeutic procedures (e.g.ERCP or colonoscopies), regular breathing is often disturbed by moving, squeezing, coughing or changes between nose and mouth ventilation causing leakage and therefore artifacts or misinterpretation of data acquired with ETCO2. These problems often restrict the use of side-stream capnography in clinical practice, although the American Society of Anesthesiologists have suggested in their guidelines that extended monitoring with capnography 'should be considered'in deep sedation. The oxygen reserve index (ORI) is a new feature of multiple wavelength pulse oximetry that provides real-time visibility to oxygenation status in the moderate hyperoxic range (PaO2 of approximately 100-200 mm Hg). The ORI is an "index" with a unit-less scale between 0.00 and 1.00 that can be trended and has optional alarms to notify clinicians of changes in a patient's oxygen status. When utilized in conjunction with SpO2 monitoring the ORI may extend the visibility of a patient's oxygen status into ranges previously unmonitored in this fashion. The ORI may make pre-oxygenation visible, may provide early warning when oxygenation deteriorates, and may facilitate a more precise setting of the required FiO2 level. In this study we aimed to show effectivity of capnography and ORİ monitoring to avoid respiratory events and hypoxia in sedated endoscopic patients. In this study we targeted totally 300 sedated endoscopy patients. Patients will randomize to two groups. In Group I anaesthesiologis will be able to use all the monitoring, where as in Group II will be blinded for ORİ. We will apply pre-oxygenation to obtain long safe apnea time. Approximately 5 min pre-oxygenation (5L/min via nasal cannula) will be used to reach steady state in oxygen reserve. We defined hypoxemia ; SpO2<95% and severe hypoxemia SpO2≤90%, hypoventilation; rise10 mmHg in ETCO2 compare to baseline, ETCO2≤30 mmHg and flat capnography.

DETAILED DESCRIPTION:
Endoscopy constitutes a wide range of procedures with many indications. Esophagogastroduodenoscopy, colonoscopy, endoscopic retrograde cholangiopancreatography (ERCP), endoscopic ultrasonography (EUS), and enteroscopy comprise the most commonly performed procedures.

There has been a considerable progress in the practice of sedation and anaesthesia for endoscopic procedures. The use of sedation reduces patient discomfort and anxiety while improving the technical quality of the procedure, and as a result, over 98% of clinicians have adopted the practice. The tremendous benefits of sedation are offset by heightened costs, increased patient discharge time, and cardiopulmonary complication risks.(1) It has been well accepted that the most important negative impact of sedation and anaesthesia is the compromise of respiratory function in the form of hypoxemia, hypoxia and alveolar hypoventilation. Recent analysis of procedural sedation has revealed an overall incidence of respiratory depression of 4,1%, with 1,1% of patients requiring assisted ventilation or reversal agents for respiratory depression.(2) Respiratory monitoring is a fundamental component of every anaesthetic regimen. Its major relevance for maintenance of homeostasis and patients' safety is recognized in its position as a mandatory element in national and international standards for anaesthetic monitoring. (3)Through the decades, advances in respiratory monitoring have reduced the incidence of anaesthetic morbidity and mortality and have opened a new era of safe anaesthetic practice. The inherent liabilities of putting patients under sedation have necessitated a large number of physiological monitoring systems in order to ensure patient comfort and safety. Currently American Society of Anaesthesiologist (ASA) guidelines recommend monitoring of pulse oximetry, blood pressure, heart rate, and end-tidal CO2; although important safeguards, these physiological measurements do not allow for the reliable assessment of patient sedation. Proper monitoring of patient state ensures procedure quality and patient safety; however no "gold-standard" is available to determine the depth of sedation, which is comparable to the anaesthesiologist's professional judgment. The 2010 House of Delegates of the American Society of Anaesthesiologists (ASA) amended its Standards for Basic Anaesthetic Monitoring to include mandatory exhaled end-tidal carbon dioxide (ETCO2) monitoring during both moderate and deep sedation to its existing requirement for endotracheal and laryngeal mask airway general anaesthesia. (4) Changes in the respiratory rate, visual inspection of the chest rise and pulse oximetry (SpO2) have been considered the most conventional and oldest non-invasive methods to determine changes in the ventilator status of patients.(5,6) However, derived respiratory rate alone cannot measure of ventilation. Clinical organization guidelines and growing body of studies suggest that respiratory rate alone is an inadequate measure of ventilation, as severe respiratory depression may develop in the presence of a normal respiratory rate.(7,8) Pulse oximetry (SpO2) is a non-invasive, reliable, and simple method for continuously monitoring the fractional arterial oxygen saturation and is essential component of respiratory monitoring. SpO2 is an estimate of SaO2 and it does not provide information about tissue oxygenation. Moreover SpO2 does not completely reflect ventilation.(9) Due to the S-shape of the oxygen dissociation curve, large changes in the partial oxygen tension (PaO2) may remain unnoticed over a period of time if monitoring is carried out with SpO2 alone.(10) If healthy subjects are pre-oxygenated with 100% oxygen and ventilate effectively and then become apneic, it may take up to 6 min for an adult before SpO2 drops below 90%. (11)

Monitoring ETCO2 for the anaesthesiologists is far superior to the pulse oximeter for immediately detecting an obstructed airway, opiate induced apnea, or other airway problems that only much later may be detected by the pulse oximeter. As hypoventilation is directly reflected by an increase in arterial carbon dioxide tension (PaCO2), capnography suggests itself as an additional monitoring parameter, which furthermore demonstrates respiration activity breath by breath. (10,12,13) Monitoring ETCO2 is particularly important when anaesthesiologists provide moderate sedation for patients who are medically compromised, such as an ASA IV patient with severe chronic obstructive pulmonary disease who may retain high levels of CO2 during sedation or a morbidly obese, insulin-dependent diabetic patient with severe obstructive sleep apnea. Additionally, in the case of colonoscopy the anaesthesiologist's only option for managing severe discomfort in the moderately sedated patients is to deepen the level of sedation until the patient becomes unconsciousness, when monitoring ETCO2 may be deemed much more important. ASA believes that other less qualified, non-anaesthesiologist sedation practitioners need it even more than anaesthesiologists.(4) Some of the independent risk factors for hypoxemia described by Friedrich-Rust et al. are age, high body mass index, history of sleep apnea, standart monitoring group (without capnography), total dose of propofol and dose of ketamine.(14) Quader et al. found a significant difference in the detection of hypoxemic events in 247 patients undergoing an endoscopic procedure using capnography versus routine surveillance. When capnography was blinded to the health care provider, 69% of the patients developed hypoxemia compared to 46% when capnography was available to the provider (p<0.001).(15) Slagelse et al. explored if the addition of capnography to standard monitoring during endoscopy could reduce number, duration and level of hypoxia in 540 patients. They found that the number and total duration of hypoxia was reduced by 39,3 and 21,1% in the intervention group compared to the control group (p>0.05). (16) Actually in intubated patients or under stable conditions without oral leakage the measurement of end-tidal carbon dioxide tension in the exhaled air shows an adequate correlation with PaCO2.(10) Unfortunately, in the state of moderate or deep sedation during diagnostic or therapeutic procedures (e.g.ERCP or colonoscopies), regular breathing is often disturbed by moving, squeezing, coughing or changes between nose and mouth ventilation causing leakage and therefore artifacts or misinterpretation of data acquired with ETCO2. These problems often restrict the use of side-stream capnography in clinical practice, although the American Society of Anesthesiologists as well as the American Society of Gastrointestinal Endoscopy (ASGE) have suggested in their guidelines that extended monitoring with capnography 'should be considered'in deep sedation. (12,17) Furthermore, while breathing room air, alveolar hypoventilation can be easily detected with capnography as an increase in the ETCO2. Since the alveolar oxygen partial pressure decreases, it may lead to an immediate decrease of SpO2. However up to 35% of all hypoxemic events in patients undergoing endoscopic procedures occur with completely normal ventilation. In contrast, supplemental oxygen results in increased alveolar oxygen partial pressure despite the presence of hypoventilation. Rising ETCO2 and/or flattening of capnography indicates hypoventilation with hypoxia being a relatively late finding, especially in a patient receiving supplemental oxygen. (18) Arakawa et al. recently evaluated the masking effects of oxygen supplementation in SpO2 when alveolar ventilation develops during sedated endoscopy in 70 patients. They found that SpO2 was significantly higher in the oxygen supplementation group than in the group breathing room air (98.6 1,4% vs 93,1 p<0.001) at peak ETCO2, and oxygen supplementation caused SpO2 to be overestimated by greater than 5% when compared with room air. SpO2 at peak ETCO2 was reduced from the baseline before sedation for the oxygen supplementation and room air breathing groups by 0,5 1,1% and 4,1 3,1% respectively (p<0.001). (19) The patients breathing a FiO2 as little as 1 L/min via nasal cannula could be at risk for extreme hypercarbia and CO2 narcosis from inadequate breathing before patient's arterial hemoglobin oxygen saturation falls below 90%. (20) Under these circumstances, it's the visual inspection of the chest that may alert the clinician on the presence of hypoventilation. Even capnography monitoring during neurosurgery has been reported by several studies as a non-reliable method to monitor CO2 due to its underestimation of the PaCO2. (6)

Masimo Corporation has developed a new parameter for noninvasive monitoring by optical sensors, Oxygen Reserve index (ORI). The oxygen reserve index (ORI) is a new feature of multiple wavelength pulse oximetry that provides real-time visibility to oxygenation status in the moderate hyperoxic range (PaO2 of approximately 100-200 mm Hg). The ORI is an "index" with a unit-less scale between 0.00 and 1.00 that can be trended and has optional alarms to notify clinicians of changes in a patient's oxygen status. When utilized in conjunction with SpO2 monitoring the ORI may extend the visibility of a patient's oxygen status into ranges previously unmonitored in this fashion. The ORI may make pre-oxygenation visible, may provide early warning when oxygenation deteriorates, and may facilitate a more precise setting of the required FiO2 level.(21) The administration of high levels of inspired O2 before tracheal intubation (pre-oxygenation) is considered to be a routine practice as oxygen reserves are not always sufficient to prevent hypoxia during the duration of intubation.(22) The ORI may make this process visible, ensuring that the PaO2 is indeed rising in the presence of a constant maximal SpO2 level. The ORI may eventually become a performance indicator, attesting to the fact that pre-oxygenation has indeed been properly performed. Monitoring the ORI may be especially important in the presence of predictive risk factors for inadequate pre-oxygenation, which overlap with criteria predictive of difficult mask ventilation.(22) It may also be extremely important during pre-oxygenation before suctioning hypoxemic patients (23), during emergency rapid sequence induction, in obese patients, during intubation in the ICU, and especially in hypoxic patients who may require non-invasive ventilation before intubation.(21) The ORI may provide early warning of impending hypoxia before any changes in SpO2 occur. In anesthetized pediatric patients the mean time (±SD) from the start of the ORI alarm to a decrease in SpO2 below 98 % and from SpO2 98 to 90 % was 40 ± 523 and 52 ± 44 s, respectively. (24) In another recent trial in 103 anesthetized adult patients, ORI could be calculated ~91.5 % of monitored time, and was positively correlated with PaO2 values ≤240 mmHg but not with PaO2 >240 mmHg. PaO2 was ≥150 mmHg in 96.5 % of ORI >0.54, and was >100 mmHg for all ORI >0.24 (25)The early warning that the ORI provides before any decrease in SpO2 occurs may provide precious time for an earlier detection of the event and the provision of timely remedial measures.(21) Most of the studies about ETCO2 monitoring in moderate and deep sedation patients focused on the range of hypoxic events with or without ETCO2 monitoring.

ELIGIBILITY:
Inclusion Criteria:

* 300 patients with age between 18-75 who are scheduled for endoscopic procedures under moderate or deep sedation, in Türkiye Yüksek İhtisas Training and Research Hospital.

Exclusion Criteria:

* 1- Patient who refuse to concent. 2- Hepatic disease, e.g. twice the normal level of liver enzymes. 3- EF<40%.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-12-25 (Actual); Primary Completion 2016-05-25 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Hypoxemia | during the procedure when/if occured
  SpO2<95%
Severe hypoxemia | during the procedure when/if occured
  SpO2≤90%,

SECONDARY OUTCOMES:
hypoventilation | during the procedure when/if occured
  rise10 mmHg in ETCO2 compare to baseline, ETCO2≤30 mmHg and flat capnography.
low oxygen reserve index | during the procedure when/if occured
  decreases 10% compare baseline in ORI level.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Merry AF, Cooper JB, Soyannwo O, Wilson IH, Eichhorn JH. International Standards for a Safe Practice of Anesthesia 2010. Can J Anaesth. 2010 Nov;57(11):1027-34. doi: 10.1007/s12630-010-9381-6. Epub 2010 Sep 21. No abstract available. PMID 20857254
- [Result] Sacchetti A, Senula G, Strickland J, Dubin R. Procedural sedation in the community emergency department: initial results of the ProSCED registry. Acad Emerg Med. 2007 Jan;14(1):41-6. doi: 10.1197/j.aem.2006.05.023. Epub 2006 Aug 31. PMID 16946280